CLINICAL TRIAL: NCT05944237
Title: A Cancer Research UK Phase I/IIa Trial of HTL0039732, Given Orally as Monotherapy and in Combination With Immunotherapy or Other Approved Therapies in Participants With Advanced Solid Tumours
Brief Title: HTL0039732 in Participants With Advanced Solid Tumours
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Collaborators: Nxera Pharma UK Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRUKD/22/001; IRAS ID: 1006164 (Other: IRAS)
Record Dates: First submitted 2023-06-26; First posted 2023-07-13 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Neoplasms; Prostatic Neoplasms, Castration-Resistant; Stomach Neoplasms; Esophageal Neoplasms; Head and Neck Neoplasms; Colorectal Neoplasms; Pancreatic Neoplasms; Lung Neoplasms; Urinary Bladder Neoplasms; Mesothelioma, Malignant; Uterine Cervical Neoplasms; Kidney Neoplasms; Sarcoma; Pheochromocytomas
Keywords: EP4 antagonist; Anti-PD-1/PD-L1 agents; PGE2; EP4; COX inhibitor
MeSH Terms: conditions — Neoplasms; Prostatic Neoplasms, Castration-Resistant; Stomach Neoplasms; Esophageal Neoplasms; Head and Neck Neoplasms; Colorectal Neoplasms; Pancreatic Neoplasms; Lung Neoplasms; Urinary Bladder Neoplasms; Mesothelioma, Malignant; Uterine Cervical Neoplasms; Kidney Neoplasms; Sarcoma; Pheochromocytoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phase 1 Part A HTL0039732 (Dose Escalation Monotherapy) (Experimental): Groups of participants will receive increasing doses of HTL0039732 Capsules as a single agent to find a safe dose and a dose that best targets cancer cells.
  Interventions: Drug: HTL0039732 Capsules
- Phase 1 Part B HTL0039732 and Atezolizumab (Dose Escalation Combination) (Experimental): Groups of participants will receive increasing doses of HTL0039732 Capsules in combination with a fixed 1200 mg dose of atezolizumab to find a RP2D for HTL0039732.
  Interventions: Drug: HTL0039732 Capsules and atezolizumab infusion
- Phase 2a HTL0039732 and Atezolizumab (Dose Expansion Combination) (Experimental): An expansion cohort will receive the RP2D of HTL0039732 Capsules in combination with a fixed 1200 mg dose of atezolizumab.
  Interventions: Drug: HTL0039732 Capsules and atezolizumab infusion

INTERVENTIONS:
Drug: HTL0039732 Capsules — HTL0039732 Capsules will be administered orally to fasted participants, although an exploration of food effects may be performed as a single dose at Cycle 0. A single dose will be administered between 3 and 9 days prior to commencement of Cycle 1. From Cycle 1 Day 1, HTL0039732 will be administered on a once daily (QD) schedule. Each administration cycle will consist of 21 days with no break between cycles. Participants may initially receive up to 18 cycles but may continue for a further 18 cycles if they are deemed to be benefitting.
  Arms: Phase 1 Part A HTL0039732 (Dose Escalation Monotherapy)
Drug: HTL0039732 Capsules and atezolizumab infusion — HTL0039732 Capsules will be administered orally on a QD schedule to participants starting on Cycle 1 Day 1. Each administration cycle will consist of 21 days with no break between cycles. Participants will also receive 1200 mg atezolizumab as an IV infusion on Day1 of each cycle (i.e. every 3 weeks). Participants may initially receive up to 18 cycles of HTL0039732 but may continue for a further 18 cycles if they are deemed to be benefitting, and they may receive up to 36 cycles of atezolizumab.
  Arms: Phase 1 Part B HTL0039732 and Atezolizumab (Dose Escalation Combination); Phase 2a HTL0039732 and Atezolizumab (Dose Expansion Combination)

SUMMARY:
The purpose of this trial is to evaluate a new drug, HTL0039732, that will be administered on its own (as a monotherapy) and in combination with atezolizumab or with other approved anti-cancer therapies, in participants with advanced solid tumours.

DETAILED DESCRIPTION:
The trial will investigate HTL0039732, a novel specific E-type prostanoid receptor 4 (EP4) antagonist, as a monotherapy and in combination with atezolizumab, a monoclonal antibody that binds to the programmed death ligand 1 (PD-L1). The trial may be expanded in future to also evaluate HTL0039732 in combination with other approved anti-cancer therapies. HTL0039732 is a small molecule drug that blocks activation of EP4 receptors by prostaglandin E2 (PGE2), a naturally occurring substance in the body.

Prostaglandin E2 may be elevated in cancer and signalling via the EP4 receptor can lead to suppression of immune activity, allowing the cancer to escape from the immune system. Blocking the EP4 receptor may relieve that immunosuppression, allowing the immune system to be active against the cancer again.

Atezolizumab is an established immune checkpoint inhibitor that overcomes a key immunosuppressive signal and improves the magnitude and quality of tumour-specific T-cell responses, resulting in improved anti-cancer activity. It, and other similar agents, are approved for the treatment of several different types of cancer. As a common mechanism of immune suppression, immune checkpoint inhibitors also have a role in combination immunotherapies and combining EP4 inhibition by HTL0039732 with PD-L1 blockade by atezolizumab, is expected to have increased activity.

The trial will investigate HTL0039732 as a monotherapy and in combination with atezolizumab, and potentially with other approved anti-cancer therapies, in participants with advanced solid tumours (Phase 1 Part A) and in participants with advanced solid tumours where PGE2/EP4 signalling is believed to be more prevalent or significant (Phase 1 Part B and Phase 2a).

This is a first-in-human clinical trial and is split as follows:

* Phase 1 is the 'dose escalation' phase, where two groups (known as Part A and Part B) of participants with solid tumours will receive increasing doses of HTL0039732 to find the safest dose.
* Part A participants will receive HTL0039732 as a single agent.
* Part B participants will receive HTL0039732 in combination with atezolizumab.
* More Parts may be added in future for participants to receive HTL0039732 in combination with other approved anti-cancer therapies.
* Phase 2a is the 'dose expansion' phase, where participants grouped according to the type of cancer they have will receive the recommended Phase 2 dose (RP2D) of HTL0039732 in combination with atezolizumab, and potentially in combination with other approved anti-cancer therapies. Phase 2a will follow a response enrichment approach; activity of the investigational medicinal products will be assessed in each group and ongoing recruitment will focus on tumour types with promising signals.

The main aims of the clinical trial are to find out:

* The most appropriate dose of HTL0039732 administered on its own, and the most appropriate dose/s of HTL0039732 to take forward for further investigation in combination with atezolizumab and with other approved anti-cancer therapies.
* More about any potential side effects of HTL0039732 when given alone and in combination with atezolizumab and other approved anti-cancer therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Written (signed and dated) informed consent and capable of co-operating with investigational medicinal product administration and follow-up.
2. Phase 1, dose escalation phase

   Part A (HTL0039732 monotherapy):
   * Histologically or cytologically proven advanced solid tumour, refractory to conventional treatment, or for which no further conventional therapy is considered appropriate by the Investigator or is declined by the potential participant.
   * At least 1 measurable lesion according to RECIST v1.1, which (in the Investigator's opinion) has had objective radiological progression on or after the last therapy, or at least one assessable lesion e.g. pleural or peritoneal thickening that does not fulfil RECIST v1.1 criteria for measurable disease.

     a. Consent for fresh tumour biopsy sample(s) at time of PD, if the participant has accessible disease and is eligible to receive atezolizumab. Optional at time of disease progression.
   * Consent to access and analysis of any available archival tissue or a fresh tumour sample at baseline, if archival tissue is unavailable.
   * Consent for fresh tumour biopsy sample(s) at time of PD, if the participant has accessible disease and is eligible to receive atezolizumab. Optional at time of disease progression.

   Phase 1 Part B:

   - Histologically proven advanced solid tumour where PGE2/EP4 signalling is believed to be more prevalent or significant (such as microsatellite stable colorectal cancer (MSS CRC), gastro-esophageal cancer, head and neck squamous cell carcinoma (HNSCC), mCRPC, pancreatic cancer, lung cancer, bladder cancer, mesothelioma, cervical cancer, renal cancer, sarcoma, pheochromocytoma and cancers with PI3K/AKT/mTOR pathway activating mutations using a clinically-validated assay).

   Phase 2a:

   - Histologically proven advanced solid tumour, in line with indications listed below, refractory to conventional treatment, or for which no conventional therapy is considered appropriate by the Investigator or is declined by the potential participant:
   1. MSS CRC with PIK3CA or HER2 mutation, and/or other driver mutation as agreed with the Sponsor (genomic alteration to have been previously identified using a validated next-generation sequencing method performed on either tumour tissue or circulating tumour DNA [ctDNA]);
   2. Gastric or gastroesophageal junction (GOJ) adenocarcinoma;
   3. Clear cell renal cell carcinoma;
   4. mCRPC

   Phase 1 Part B and Phase 2a:
   * Consent to access and analysis of any available archival tissue.
   * Consent for fresh tumour biopsy samples at baseline and on treatment. However, the following exceptions will be permitted if archival tissue is available at the recruiting site:

     1. Patients with mCRPC: biopsies are not required for those whose only safely accessible lesions are bone metastases that lack an accessible soft tissue component.
     2. For the first 12 participants in each indication: the on-trial biopsy is optional; and the baseline biopsy is mandatory if there is a safely accessible lesion but may be omitted for patients who have no safely accessible lesion, to permit their inclusion in the study. This will continually be assessed through the study.
   * Disease refractory to conventional treatment, or for which no further conventional therapy is considered appropriate by the Investigator or is declined by the participant.
   * Except for mCRPC, at least 1 measurable lesion according to RECIST v1.1, which (in the Investigator's opinion) has had objective radiological progression on or after the last therapy. Potential participants with mCRPC may instead have had PD according to PCWG3 criteria.

     1. Previously irradiated lesions cannot be counted as target lesions unless clearly progressed after the radiotherapy.
     2. Lesions that are intended to be biopsied should not be counted as target lesions (those undergoing biopsy must have at least one target lesion that is not intended to be biopsied).
   * For indications where anti-PD-1/PD-L1 therapy is standard of care (such as clear cell renal cell carcinoma, or gastric or GOJ adenocarcinoma with elevated PD-L1 expression), patients must have received that therapy and must be considered to have had progressive disease by the Investigator either on, or within 6 months after, that treatment.
3. Life expectancy of at least 12 weeks.
4. Eastern Cooperative Oncology Group performance status of 0 or 1.
5. Haematological and biochemical indices within the protocol specified ranges.
6. Stable thyroid function tests. Stable doses of thyroxine replacement are permitted.
7. Aged 18 years or over at the time consent is given.

Exclusion Criteria:

1. Radiotherapy (except for palliative reasons), chemotherapy, non chemotherapy systemic anti-cancer therapy (apart from life-long hormone suppression such as luteinising hormone-releasing agents in participants with mCRPC) or investigational medicinal products during the 4 weeks prior to enrolment; or first dose of an immunotherapy during the previous 12 weeks before first dose of HTL0039732.
2. Ongoing toxic manifestations of previous treatments that are Grade >1 per CTCAE v5.0.
3. Any central nervous system metastases (unless potential participants have had local therapy and are asymptomatic, radiologically stable and have been off steroids for ≥4 weeks prior to enrolment).
4. Women of child-bearing potential (or who are already pregnant or lactating). Exceptions apply.
5. Men with partners of childbearing potential. Exceptions apply.
6. Major thoracic or abdominal surgery from which the potential participant has not yet recovered.
7. At high medical risk because of non-malignant systemic disease, including active uncontrolled infection.
8. Known history of current or latent tuberculosis, HIV or Hepatitis B or C infection.
9. Prior treatment with EP4 inhibitor.
10. Treatment with selective cyclooxygenase-2 inhibitor in the 8 weeks prior to enrolment.
11. Known hypersensitivity or intolerance to hydroxypropyl methylcellulose.
12. Use of systemic immunosuppressive agent in the 2 weeks prior to enrolment. Exceptions apply.
13. Significant cardiovascular disease.
14. Known active peptic ulcer disease, or symptoms of gastritis, dyspepsia or gastro-esophageal reflux disease (one or more episodes per week).
15. Current or planned participation in another interventional clinical trial, whilst taking part in this trial of HTL0039732.
16. Limited ability to swallow or absorb oral medications.
17. Any other condition that, in the Investigator's opinion, would mean that the trial is not in the best interests of the potential participant.

    Phase 1 Part B and Phase 2a:
18. Any live vaccines in the 4 weeks prior to enrolment.
19. Diagnosis of immunodeficiency.
20. Active autoimmune disease requiring systemic treatment in the 2 years prior to enrolment.
21. History or clinical suspicion of interstitial lung disease, history of (non-infectious) pneumonitis that required steroids, or current pneumonitis.
22. Hypersensitivity to atezolizumab or any of its excipients.
23. Prior adverse reaction to cancer immunotherapy that required steroid or other immunosuppressive treatment or led to discontinuation of that treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-07-13 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD; Dose Escalation Phase) | From first dose of HTL0039732 up to the end of Cycle 1, a time frame of up to 30 days.
  The MTD is the highest dose of HTL0039732 in the safe dose range, i.e. where there is a <25% probability of toxicity being above 30%.
RP2D (Dose Escalation Phase) | From first dose of HTL0039732 up to the off-study visit (maximum 115 weeks).
  The RP2D for HTL0039732 will be determined after reviewing all of the clinically relevant toxicity, efficacy and pharmacokinetic (PK)/pharmacodynamic data by the Trial Management Group.
Number of Adverse Events (AEs) Related to HTL0039732 (Dose Escalation and Expansion Phase) | Safety data will be collected from the time of informed consent until 28 days after the last dose of HTL0039732. The average time from consent to the end of follow-up will be presented.
  Number of all grade AEs, and number of Grade 3, 4 and 5 AEs, considered at least possibly related to HTL0039732, graded according to National Cancer Institute Common Criteria for Adverse Events (NCI CTCAE) Version 5.0. Count of AEs by arm.
Number of AEs Related to Atezolizumab (Dose Escalation and Expansion Phase) | Safety data will be collected from the time of informed consent until 90 days after the last dose of atezolizumab. The average time from consent to the end of follow-up will be presented.
  Number of all grade AEs, and number of Grade 3, 4 and 5 AEs, considered at least possibly related to atezolizumab, graded according to NCI CTCAE Version 5.0. Count of AEs by arm.

SECONDARY OUTCOMES:
Measurement of the PK Parameter Maximum (or Peak) Plasma Concentration (Cmax) of HTL0039732 (Dose Escalation and Expansion Phase) | From first dose of HTL0039732 until Cycle 6 Day 1 (max. 20 weeks).
  Plasma samples will be analysed by liquid chromatography with tandem mass spectrometry (LC-MS/MS) to determine the Cmax of HTL0039732 after oral administration of HTL0039732 Capsules as monotherapy and in combination with atezolizumab, according to agreed standard operating procedures (SOPs) and validated methods. Not all participants may be analysed at all time points.
Measurement of the PK Parameter Time to Reach Maximum (or Peak) Plasma Concentration (Tmax) of HTL0039732 (Dose Escalation and Expansion Phase) | Timeframe: From first dose of HTL0039732 until Cycle 6 Day 1 (max. 20 weeks).
  Plasma samples will be analysed by LC-MS/MS to determine the Tmax of HTL0039732 after oral administration of HTL0039732 Capsules as monotherapy and in combination with atezolizumab, according to agreed SOPs and validated methods. Not all participants may be analysed at all time points.
Measurement of the PK Parameter Minimum Plasma Concentration (Cmin) of HTL0039732 (Dose Escalation and Expansion Phase) | From first dose of HTL0039732 until Cycle 6 Day 1 (max. 20 weeks).
  Plasma samples will be analysed by LC-MS/MS to determine the Cmin of HTL0039732 after oral administration of HTL0039732 Capsules as monotherapy and in combination with atezolizumab, according to agreed SOPs and validated methods. Not all participants may be analysed at all time points.
Measurement of the PK Parameter Area under the Plasma Concentration-Time Curve (AUC) (Dose Escalation and Expansion Phase) | From first dose of HTL0039732 until Cycle 6 Day 1 (max. 20 weeks).
  Plasma samples will be analysed by LC-MS/MS to determine the AUC of HTL0039732 after oral administration of HTL0039732 Capsules as monotherapy and in combination with atezolizumab, according to agreed SOPs and validated methods. Not all participants may be analysed at all time points.
Measurement of the PK Parameter Apparent Clearance (CL/F) (Dose Escalation and Expansion Phase) | From first dose of HTL0039732 until Cycle 6 Day 1 (max. 20 weeks).
  Plasma samples will be analysed by LC-MS/MS to determine the CL/F of HTL0039732 after oral administration of HTL0039732 Capsules as monotherapy and in combination with atezolizumab, according to agreed SOPs and validated methods. Not all participants may be analysed at all time points.
Measurement of the PK Parameter Apparent Volume of Distribution (V/F) (Dose Escalation and Expansion Phase) | From first dose of HTL0039732 until Cycle 6 Day 1 (max. 20 weeks).
  Plasma samples will be analysed by LC-MS/MS to determine the V/F of HTL0039732 after oral administration of HTL0039732 Capsules as monotherapy and in combination with atezolizumab, according to agreed SOPs and validated methods. Not all participants may be analysed at all time points.
Measurement of the PK Parameter Terminal Elimination Half-Life (T1/2) (Dose Escalation and Expansion Phase) | From first dose of HTL0039732 until Cycle 6 Day 1 (max. 20 weeks).
  Plasma samples will be analysed by LC-MS/MS to determine the T1/2 of HTL0039732 after oral administration of HTL0039732 Capsules as monotherapy and in combination with atezolizumab, according to agreed SOPs and validated methods. Not all participants may be analysed at all time points.
Determine the magnitude and duration of de-repression of inhibition by prostaglandin E2 of lipopolysaccharide induced tumour necrosis alpha production, ex vivo in whole blood | From first dose of HTL0039732 until Cycle 2 Day 8 (max. 6 weeks).
  Mean percentage reversal at timepoints from baseline to final timepoint.
Best Anti-Tumour Response to HTL0039732 According to Response Evaluation Criteria in Solid Tumours (RECIST) version (v) 1.1 (Dose Escalation Phase Part A) | From baseline radiological disease assessment until End of Study visit (max. 118 weeks). Efficacy follow-up may continue until end of trial.
  Best radiological response, presented per arm by count of participants: complete response (CR), partial response (PR), stable disease (SD) or progressive disease (PD), based on RECIST v1.1. A CR or PR should be confirmed by a subsequent assessment ≥4 weeks later. SD criteria must be met at least once ≥6 weeks after trial entry to be defined as SD.
Best Overall Response to HTL0039732 and Atezolizumab According to RECIST v 1.1 or Prostate Cancer Clinical Trials Working Group 3 (PCWG3) (Dose Escalation Phase Part B and Dose Expansion Phase) | From baseline radiological disease assessment until End of Study visit (max. 118 weeks). Efficacy follow-up may continue until end of trial.
  Best radiological response, presented per arm by count of participants: CR, PR, SD or PD, based on RECIST v1.1, or based on PCWG3 for participants with prostate cancer. For a participant to have a CR or PR, the response needs to be confirmed by a subsequent assessment ≥4 weeks later. SD criteria must be met at least once ≥6 weeks after trial entry to be defined as SD.
Objective Response Rate according to RECIST 1.1 or by PCWG3 criteria (Dose Escalation Phase Part B and Dose Expansion Phase) | From baseline radiological disease assessment until End of Study visit (max. 118 weeks). Efficacy follow-up may continue until end of trial.
  Percentage of participants, presented per arm, with CR or PR, based on RECIST v1.1, or based on PCWG3 for participants with prostate cancer. For a participant to have a CR or PR, the response needs to be confirmed by a subsequent assessment ≥4 weeks later.
Duration of Response according to RECIST 1.1 or by PCWG3 criteria (Dose Escalation Phase Part B and Dose Expansion Phase) | From time of first response until End of Study visit (max. 118 weeks). Efficacy follow-up may continue until end of trial.
  The time in days from the date of first response (defined as CR or PR) to the date when PD is first identified, based on RECIST v1.1, or based on PCWG3 for participants with prostate cancer. For a participant to have a CR or PR, the response needs to be confirmed by a subsequent assessment ≥4 weeks later.
Disease Control Rate according to RECIST 1.1 or by PCWG3 criteria (Dose Escalation Phase Part B and Dose Expansion Phase) | From baseline radiological disease assessment until End of Study visit (max. 118 weeks). Efficacy follow-up may continue until end of trial.
  Percentage of participants, presented per arm, with CR, PR or SD, based on RECIST v1.1, or based on PCWG3 for participants with prostate cancer. For a participant to have a CR or PR, the response needs to be confirmed by a subsequent assessment ≥4 weeks later. SD criteria must be met at least once ≥6 weeks after trial entry to be defined as SD.
Progression Free Survival according to RECIST 1.1 or by PCWG3 criteria (Dose Escalation Phase Part B and Dose Expansion Phase) | From first dose of HTL0039732 until End of Study visit (max. 118 weeks). Efficacy follow-up may continue until end of trial.
  The time in days from first dose of HTL0039732 until the time at which PD is identified, based on RECIST v1.1, or based on PCWG3 for participants with prostate cancer. For a participant to have a CR or PR, the response needs to be confirmed by a subsequent assessment ≥4 weeks later. SD criteria must be met at least once ≥6 weeks after trial entry to be defined as SD.
Prostate Specific Antigen (PSA) response of at least 50% for participants with metastatic castration resistant prostate cancer (mCRPC) (Dose Escalation Phase Part B and Dose Expansion Phase) | At least 12 weeks after baseline PSA.
  Percentage of participants with mCRPC showing a reduction from baseline in PSA response ≥50%.
Change in sum of target lesions according to RECIST 1.1 or by PCWG3 criteria (Dose Escalation and Dose Expansion Phase). | From baseline radiological disease assessment until End of Study visit (max. 118 weeks).
  The change in the sum of diameters (SOD) for all target lesions calculated (by using the longest diameter for soft-tissue lesions and short axis for nodal lesions) will be reported.
Assess tumour T cell infiltration in baseline and on-treatment biopsies | Baseline to Cycle 1 Day 15 (±7 days).
  CD8 positive T-cells at baseline and on-treatment (biopsy).
Assess change in tumour T cell infiltration in baseline and on-treatment biopsies | Baseline to Cycle 1 Day 15 (±7 days).
  Fold change in CD8 positive T-cells between baseline and on-treatment biopsy.

CONTACTS AND LOCATIONS:
Locations (5):
- United Kingdom (5):
  - Addenbrooke's Hospital, Cambridge
  - Velindre Cancer Centre, Cardiff
  - Clatterbridge Cancer Centre, Liverpool
  - Guy's Hospital, London
  - The Christie Hospital, Manchester

IPD SHARING:
Plan to Share IPD: No